CLINICAL TRIAL: NCT05296473
Title: Guided ADHD Therapy for Managing the Extent and Severity of Symptoms - A Randomized, Controlled, Parallel-group, Intervention Study to Assess an At-home, Game-based Digital Therapy for Treating Adult Patients With Attention-Deficit/Hyperactivity Disorder
Brief Title: Guided ADHD Therapy for Managing the Extent and Severity of Symptoms
Acronym: GAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIP-013
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD Therapy (Experimental)
  Interventions: Device: ADHD Therapy
- Control Therapy (Active Comparator)
  Interventions: Device: Control Therapy

INTERVENTIONS:
Device: ADHD Therapy — investigational game-play therapy
  Arms: ADHD Therapy
Device: Control Therapy — control game-play therapy
  Arms: Control Therapy

SUMMARY:
The objective of this study is to assess the safety and effectiveness of an at-home, game-based digital therapy for treating adult patients with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects 22-55 years of age
* Male or female
* Confirmed ADHD diagnosis, combined or inattentive type, at Screening based on DSM-5 criteria and established via the MINI-Adult, administered by a trained clinician
* Baseline score on the clinician-rated ADHD-RS total score ≥28
* Not undergoing pharmacological treatment with methylphenidate or amphetamine-based products at time of Screening; or, if undergoing pharmacological treatment, must be willing and appropriate (i.e., not optimally treated in the Investigator's judgement or having issues with tolerability) to wash out of current regimen
* Estimated IQ score ≥80 as assessed by the Kaufmann Brief Intelligence Test, Second Edition (KBIT-II)
* Ability to understand and speak English, follow written and verbal instructions (English), as assessed by the PI and/or Study Coordinator, and give informed consent (English)
* Have ability to connect wireless devices to a functional wireless network on a daily basis
* Ability to comply with all the testing and study requirements

Exclusion Criteria:

* Current, controlled (requiring restricted medication) or uncontrolled, comorbid psychiatric diagnosis, based on MINI-Adult and subsequent clinical interviewing, with significant symptoms including but not limited to posttraumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments.
* Patients who are currently treated with a non-stimulant medication for ADHD (i.e., atomoxetine, clonidine, guanfacine, viloxazine)
* Have previously been assessed by TOVA for potential enrollment in a clinical trial.
* Have previously used a videogame-like digital therapy (e.g., Akili EndeavorRxTM) OR Within the last three years, have used a cognitive or brain training platform (e.g., Peak, Brain HQ, Lumosity, Atentiv) for more than two weeks duration
* Known sensitivity to playing video games, such as headaches, dizziness, nausea.
* Initiation within the last 4 weeks of behavioral therapy or neurofeedback, or planned initiation during the study. Patients who have been in behavior therapy or neurofeedback consistently for more than 4 weeks may participate provided their routine is unchanged during the course of the study. Patients planning on changing or initiating behavior therapy or neurofeedback during the course of the study will be excluded.
* Patient is currently considered a suicide risk in the opinion of the Investigator, as measured by C-SSRS at screening (i.e., score of 4 or 5 on C-SSRS)
* Motor condition (e.g., physical deformity of the hands/arms; protheses) that prevents game playing as observed by the Investigator
* Recent history (within the past 12 months) of suspected alcohol or substance abuse or dependence
* Positive urine drug screen
* History of seizures (excluding febrile seizures), or significant motor or vocal tics, including but not limited to Tourette's Disorder and photo-sensitive epilepsy
* Visual acuity that cannot be corrected that prevents or negatively impacts game playing as observed by the Investigator
* Any use of psychoactive drugs (other than stimulant) that in the opinion of the Investigator may confound study data/assessments
* Has participated in a clinical trial within 90 days prior to screening
* Has a family member or close friend/associate also enrolled/currently participating in the same study
* Any other condition that in the opinion of the Investigator may confound study data/assessments

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 560 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Test of Variables of Attention (TOVA®) Attention Comparison Score (ACS) | Study Day 0 to Study Day 63
  The TOVA is a standardized, computerized, continuous performance test (CPT). The TOVA Attention Comparison Score (ACS) is a comparison of a subject's scores to scores from a normative ADHD population. A score of < 0 indicates a subject's performance is similar to that of the normative ADHD population, with a lower score indicating a more severe ADHD profile. A positive change on the TOVA ACS from Day 0 to Day 63 indicates improvement.

SECONDARY OUTCOMES:
ADHD-RS-5 Inattention Subscale with Adult Prompts | Study Day 0 to Study Day 63
  The ADHD-RS-5 with Adult Prompts is an 18-item, clinician-administered questionnaire that rates the frequency of occurrence of ADHD symptoms and behaviors as defined by criteria outlined for ADHD in the DSM-5. Each item is scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms). The first 9 items assess inattention symptoms and the last 9 items assess hyperactive-impulsive symptoms. Each subscale produces a sub-scale score ranging from 0-27. A higher subscale score indicates more severe ADHD symptoms and behaviors. A negative change on the inattention subscale from Day 0 to Day 63 indicates improvement.
Cambridge Brain Sciences Token Search | Study Day 0 to Study Day 63
  Token Search is a computerized task designed to assess working memory. In Token Search, subjects identify the location of a hidden token in a set of boxes while remembering where previous tokens have been found. Correctly finding a token in every box will increase difficulty level in the form of a new puzzle with an increased number of boxes. Performance is indicated by the average number of tokens found. A positive change in score on the Token Search task from Day 0 to Day 63 indicates improvement.
Cambridge Brain Sciences Spatial Span | Study Day 0 to Study Day 63
  Spatial Span is a computerized task designed to assess spatial short-term memory and based on the Corsi Block tapping task. In Spatial Span, subjects are shown a sequence of flashing boxes and have to repeat the sequence. Sequence lengths increase with correct answers. Performance is indicated by the average number of boxes remembered during the task. A positive change in score on the Spatial Span ask from Day 0 to Day 63 indicates improvement.
Behavior Rating Inventory of Executive Function - Adult Version (BRIEF-A) Working Memory and Inhibit Percentiles | Study Day 0 to Study Day 63
  The BRIEF-A is composed of 75 items within nine non-overlapping theoretically and empirically derived clinical scales that measure various aspects of executive functioning. Each item is rated as either 1 (never), 2 (sometimes), or 3 (often). A reduction in score from Day 0 to Day 63 indicates improvement.
Weiss Functional Impairment Rating Scale - Self-Report (WFIRS-S) | Study Day 0 to Study Day 63
  The WFIRS-S is a validated rating scale used to capture functional difficulties in the lives of individuals with ADHD in 7 domains. Each item is scored on a 4-point scale ranging from 0 (Never or not at all) to 3 (Very often of very much). A reduction in score from Day 0 to Day 63 indicates improvement.
Clinical Global Impression Scale - Improvement (CGI-I) | at Study Day 63
  The Clinical Global Impression Scale-Improvement (CGI-I) is a clinician's comparison of the participant's overall clinical condition at follow-up to the overall clinical condition at baseline. The CGI-I consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). A score of 1 (very much improved) or 2 (much improved) or 3 (minimally improved) would indicate overall improvement of ADHD severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Clinical Research of Southern Nevada, LLC
Locations (13):
- United States (13):
  - Melmed Center, Scottsdale, Arizona
  - CNS Network, Garden Grove, California
  - University of California Davis MIND Institute, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Accel Research Sites - Maitland Clinical Research Unit, Maitland, Florida
  - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center of Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Duke University, Durham, North Carolina
  - Mindpath Care Centers, Raleigh, North Carolina
  - CNS Healthcare, Memphis, Tennessee
  - FutureSearch Trials of Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No